CLINICAL TRIAL: NCT02701517
Title: Randomized Trial of Cyclosporine + CAMPATH-1H (ALEMTUZUMAB) vs. Cyclosporine + METHOTREXATE in Patients Diagnosed With Mature B-cell Neoplasms - Chronic Lymphocytic Leukemia and Low-grade Lymphomas - Receiving Allogeneic Hematopoietic Stem Cell Transplantation With Nonmyeloablative Conditioning Regimen
Brief Title: Cyclosporine Plus Methotrexate or Alemtuzumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped before the targeted number of patients was reached due to lack of support.
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIRCAMPATH-alo 2002
Record Dates: First submitted 2015-03-12; First posted 2016-03-08 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Unrecognized Condition: Mature B or T-cell Neoplasm
Keywords: conditioning treatment; alemtuzumab; allogeneic hematopoietic stem cell transplantation; chronic lymphoproliferative disorders
MeSH Terms: interventions — Cyclosporine; Methotrexate; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine + METHOTREXATE (Active Comparator): MTX days +1, +3, +6 and +11 followed by folinic acid rescue. All patients will receive CSA from day -7.
  Interventions: Drug: Cyclosporine + METHOTREXATE
- Cyclosporine + CAMPATH-1H (Experimental): CAMPATH-1H at a dose of 20 mg / day at 8-hour intravenous infusion on days -8 to -4. All patients will receive CSA from day -7.
  Interventions: Drug: Cyclosporine + CAMPATH-1H

INTERVENTIONS:
Drug: Cyclosporine + METHOTREXATE — MTX days +1, +3, +6 and +11 followed by rescue with folinic Ac. All patients receive CSA from day -7.
  Arms: Cyclosporine + METHOTREXATE
Drug: Cyclosporine + CAMPATH-1H — CAMPATH-1H at a dose of 20 mg / day at 8-hour intravenous infusion on days -8 to -4. All patients will receive CSA from day -7.
  Other Names: Alemtuzumab
  Arms: Cyclosporine + CAMPATH-1H

SUMMARY:
The primary aim of the study was to compare the efficacy of the procedure in terms of event-free survival between patients receiving cyclosporine (CsA) plus either alemtuzumab (CAMPATH-1H ) or methotrexate (MTX) after matched related donor allo-reduced intensity conditioning. Secondary aims were: 1. To compare the incidence of infections and transplant-related mortality between the two arms; 2. to compare the incidence of acute and chronic GVHD 3. to evaluate hematologic and immunologic reconstitution and evolution of chimerism and residual disease.

Patients were randomly assigned to received cyclosporine plus alemtuzumab or cyclosporine plus MTX and were stratified according to diagnosis: Chronic lymphocytic leukemia or Low grade- non-Hodgkin's lymphoma.

All patients received the same reduced-intensity conditioning (RIC) scheme based on fludarabine 150mg/m2 (30 mg/m2/day everyday from -8 to -4) plus melphalan 140mg/m2 (70 mg/m2/day everyday from -3 to -2). Regarding the GVHD prophylaxis, patients in group 1 (n=17) received CsA 1 mg/kg intravenously starting on day -7 and 2/mg/Kg from day -1 plus alemtuzumab administered at a dose of 20 mg IV on -8 to -4 whereas in group 2 (n=23) pts received CsA at same doses as group 1 plus MTX given at a dose of 15 mg/m2 intravenously on days 1 and 10 mg/m2 on days 3, 6 and 11, followed by folinic acid rescue (15 mg in +1 and 10 mg in +3, +6 and +11 intravenously every 6 hours for 4 doses starting 24 hours after each dose of MTX).

Acute and chronic GVHD were similarly graded by established criteria [20, 21]. In patients receiving alemtuzumab, CsA was suspended by day +130. They also received donor lymphocyte infusion (DLI) at a dose of 1 x 107 cluster of differentiation 3 / kg on day +180 in case of active disease, persistence of minimal residual disease detected by flow cytometry or mixed chimerism and no GVHD. In case mixed chimerism, donor lymphocyte infusion was performed if patient hematopoiesis progressively increased. In patients receiving CsA + MTX, CsA was suspended by day +180. These patients received DLI only in situations specified above.

The statistical analysis has been designed to identify a 20% difference in terms of disease-free survival (based on the increased incidence of relapse in patients receiving T-cell depletion).

ELIGIBILITY:
Inclusion criteria:

1. Having an identical Human Leukocyte Antigens (HLA) or a mismatched family donor.
2. Age between 45 and 65 years (outside this age range at the discretion of each center).
3. Indications:

   * Follicular lymphoma with one of the following characteristics:

     1. Poor prognosis follicular NHL (3 or more factors by Federico et al: erythrocyte sedimentation rate (ESR)> 30, male,> 60 years, high LDH> 2 extranodal areas, pathologic stage (PS) >2 or The International Prognostic Index (IPI) 3 or high lactate dehydrogenase (LDH) or micro Beta 2) failing to achieve CR with regimens including fludarabine and anti CD20 (cluster of differentiation antigen 20 ).
     2. 2nd CR (complete response) or PR (partial response) not candidates for autologous transplantation;
     3. persistent disease or relapse after autologous transplantation.
   * Other low-grade lymphomas:

     1. relapsed after autologous transplantation.
     2. autologous transplant candidates which can not be performed because of the inability to collect a sufficient number of cells, steam cells disease persistence, etc..
   * Chronic lymphocytic leukemia with one of the following characteristics:

     1. "B" symptoms: weight loss >10% in the last 6 months, fever >38ºC (degrees centigrade) for 14 days without infection, night sweats without infection
     2. lymphadenopathy >10 cm or progressive, progressive splenomegaly
     3. Anemia and/or thrombocytopenia secondary to bone marrow infiltration
     4. Diffuse lymphocytic infiltration of the bone marrow
     5. Progressive lymphocytosis (>50% in 2 months) or a lymphocyte doubling time <12 months Any of the above criteria is an inclusion criteria in the protocol in patients who have received at least one line of treatment including fludarabine
     6. Patients with poor prognostic cytogenetic abnormalities: 17p-, 11q-with VDJ unmutated
4. Patients must also meet the following general requirements:

   1. Performance status <3 (Zubrod score, Eastern Cooperative Oncology Group (ECOG) performance status or WHO (World Health Organization) )
   2. forced expiratory volume at one second (FEV1) > 39%, lung diffusing capacity for carbon monoxide (DLCO) and forced vital capacity (FVC) > 39% of the theoretical values
   3. Total bilirubin and transaminases <3 x the normal maximum value, unless attributable to base haemopathy
   4. Creatinine <2 x normal maximum and clearance> 40 mL / min unless attributable to his base haemopathy
   5. No evidence of symptomatic disease, cirrhosis or active hepatitis
   6. Negative serology for HIV
   7. Written informed consent

Exclusion criteria:

1. Impaired hepatic or renal function superior to that described above
2. Presence of serious diseases that prevent chemotherapy treatments
3. Presence of psychiatric comorbidity
4. HIV infection
5. Other prior neoplasm
6. Do not have signed informed consent
7. Pregnant or at risk of pregnancy by inadequate contraceptive measures.
8. Patients diagnosed with chronic lymphocytic leukemia (CLL) transformation to more aggressive cytologic or histologic forms (prolymphocytic leukemia, large cell lymphoma, Hodgkin's disease) and those affected with autoimmune hemolytic anemia

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2003-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of transplantation in terms of event-free survival | From +270 days
  To compare the efficacy of transplantation in terms of event-free survival between patients receiving CAMPATH-1H or methotrexate in allogeneic related donor with nonmyeloablative conditioning.

SECONDARY OUTCOMES:
Incidence of infections and transplant-related mortality | 1 year
  Compare the incidence of infections and transplant-related mortality between the two arms

OTHER OUTCOMES:
incidence of graft versus host disease | 5 years
  Analyze the impact on the incidence of graft versus host disease (GVHD) acute and chronic CAMPATH-1H + DLI compared with MTX as GVHD prophylaxis in allogeneic related donor with nonmyeloablative conditioning.

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Pérez-Simón, MD, PhD, Principal Investigator — University of Salamanca
Locations (5):
- Department of Propedeutic Oncology, Medical University of Gdansk, Gdansk, Poland
- Spain (4):
  - Clinical Hematology Department. ICO-Hospital Germans Trias i Pujol. Jose Carreras Research Institute, Badalona, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Santa Creu I Sant Pau Hospital, Barcelona
  - Hospital Universitario de Salamanca, Salamanca

REFERENCES:
- [Background] Kroger N, Shaw B, Iacobelli S, Zabelina T, Peggs K, Shimoni A, Nagler A, Binder T, Eiermann T, Madrigal A, Schwerdtfeger R, Kiehl M, Sayer HG, Beyer J, Bornhauser M, Ayuk F, Zander AR, Marks DI; Clinical Trial Committee of the British Society of Blood and Marrow Transplantation and the German Cooperative Transplant Group. Comparison between antithymocyte globulin and alemtuzumab and the possible impact of KIR-ligand mismatch after dose-reduced conditioning and unrelated stem cell transplantation in patients with multiple myeloma. Br J Haematol. 2005 Jun;129(5):631-43. doi: 10.1111/j.1365-2141.2005.05513.x. PMID 15916686
- [Background] Chen PM, Tzeng CH, Fan FS, Hsieh RK, Wei CH. Bone marrow transplantation in Taiwan: low incidence of acute GVHD in patients with hematologic malignancies and severe aplastic anemia. Bone Marrow Transplant. 1994 Jun;13(6):709-11. PMID 7920299
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Sullivan KM, Shulman HM, Storb R, Weiden PL, Witherspoon RP, McDonald GB, Schubert MM, Atkinson K, Thomas ED. Chronic graft-versus-host disease in 52 patients: adverse natural course and successful treatment with combination immunosuppression. Blood. 1981 Feb;57(2):267-76. PMID 7004534
- [Background] Morris E, Thomson K, Craddock C, Mahendra P, Milligan D, Cook G, Smith GM, Parker A, Schey S, Chopra R, Hatton C, Tighe J, Hunter A, Peggs K, Linch D, Goldstone A, Mackinnon S. Outcomes after alemtuzumab-containing reduced-intensity allogeneic transplantation regimen for relapsed and refractory non-Hodgkin lymphoma. Blood. 2004 Dec 15;104(13):3865-71. doi: 10.1182/blood-2004-03-1105. Epub 2004 Aug 10. PMID 15304395
- [Background] Delgado J, Pillai S, Benjamin R, Caballero D, Martino R, Nathwani A, Lovell R, Thomson K, Perez-Simon JA, Sureda A, Kottaridis P, Vazquez L, Peggs K, Sierra J, Milligan D, Mackinnon S. The effect of in vivo T cell depletion with alemtuzumab on reduced-intensity allogeneic hematopoietic cell transplantation for chronic lymphocytic leukemia. Biol Blood Marrow Transplant. 2008 Nov;14(11):1288-97. doi: 10.1016/j.bbmt.2008.09.001. PMID 18940684
- [Background] Perez-Simon JA, Kottaridis PD, Martino R, Craddock C, Caballero D, Chopra R, Garcia-Conde J, Milligan DW, Schey S, Urbano-Ispizua A, Parker A, Leon A, Yong K, Sureda A, Hunter A, Sierra J, Goldstone AH, Linch DC, San Miguel JF, Mackinnon S; Spanish and United Kingdom Collaborative Groups for Nonmyeloablative Transplantation. Nonmyeloablative transplantation with or without alemtuzumab: comparison between 2 prospective studies in patients with lymphoproliferative disorders. Blood. 2002 Nov 1;100(9):3121-7. doi: 10.1182/blood-2002-03-0701. PMID 12384408
- [Background] Martino R, Caballero MD, Canals C, Simon JA, Solano C, Urbano-Ispizua A, Bargay J, Rayon C, Leon A, Sarra J, Odriozola J, Conde JG, Sierra J, San Miguel J; ALLOPBSCT Subcommittee of the Spanish Group for Haematopoietic Transplantation (GETH); Group GEL-TAMO. Allogeneic peripheral blood stem cell transplantation with reduced-intensity conditioning: results of a prospective multicentre study. Br J Haematol. 2001 Dec;115(3):653-9. doi: 10.1046/j.1365-2141.2001.03153.x. PMID 11736950
- [Background] Schweighofer CD, Ritgen M, Eichhorst BF, Busch R, Abenhardt W, Kneba M, Hallek M, Wendtner CM. Consolidation with alemtuzumab improves progression-free survival in patients with chronic lymphocytic leukaemia (CLL) in first remission: long-term follow-up of a randomized phase III trial of the German CLL Study Group (GCLLSG). Br J Haematol. 2009 Jan;144(1):95-8. doi: 10.1111/j.1365-2141.2008.07394.x. Epub 2008 Oct 30. PMID 19016732
- [Background] Keating MJ, Flinn I, Jain V, Binet JL, Hillmen P, Byrd J, Albitar M, Brettman L, Santabarbara P, Wacker B, Rai KR. Therapeutic role of alemtuzumab (Campath-1H) in patients who have failed fludarabine: results of a large international study. Blood. 2002 May 15;99(10):3554-61. doi: 10.1182/blood.v99.10.3554. PMID 11986207
- [Background] Rai KR, Freter CE, Mercier RJ, Cooper MR, Mitchell BS, Stadtmauer EA, Santabarbara P, Wacker B, Brettman L. Alemtuzumab in previously treated chronic lymphocytic leukemia patients who also had received fludarabine. J Clin Oncol. 2002 Sep 15;20(18):3891-7. doi: 10.1200/JCO.2002.06.119. PMID 12228210
- [Background] Osterborg A, Dyer MJ, Bunjes D, Pangalis GA, Bastion Y, Catovsky D, Mellstedt H. Phase II multicenter study of human CD52 antibody in previously treated chronic lymphocytic leukemia. European Study Group of CAMPATH-1H Treatment in Chronic Lymphocytic Leukemia. J Clin Oncol. 1997 Apr;15(4):1567-74. doi: 10.1200/JCO.1997.15.4.1567. PMID 9193354
- [Background] Chakrabarti S, Mackinnon S, Chopra R, Kottaridis PD, Peggs K, O'Gorman P, Chakraverty R, Marshall T, Osman H, Mahendra P, Craddock C, Waldmann H, Hale G, Fegan CD, Yong K, Goldstone AH, Linch DC, Milligan DW. High incidence of cytomegalovirus infection after nonmyeloablative stem cell transplantation: potential role of Campath-1H in delaying immune reconstitution. Blood. 2002 Jun 15;99(12):4357-63. doi: 10.1182/blood.v99.12.4357. PMID 12036862
- [Background] Hale G, Cobbold S, Novitzky N, Bunjes D, Willemze R, Prentice HG, Milligan D, MacKinnon S, Waldmann H; CAMPATH Users. CAMPATH-1 antibodies in stem-cell transplantation. Cytotherapy. 2001;3(3):145-64. doi: 10.1080/146532401753173981. PMID 12171722
- [Background] Kottaridis PD, Milligan DW, Chopra R, Chakraverty RK, Chakrabarti S, Robinson S, Peggs K, Verfuerth S, Pettengell R, Marsh JC, Schey S, Mahendra P, Morgan GJ, Hale G, Waldmann H, de Elvira MC, Williams CD, Devereux S, Linch DC, Goldstone AH, Mackinnon S. In vivo CAMPATH-1H prevents graft-versus-host disease following nonmyeloablative stem cell transplantation. Blood. 2000 Oct 1;96(7):2419-25. PMID 11001893
- [Background] Khouri IF, Przepiorka D, van Besien K, O'Brien S, Palmer JL, Lerner S, Mehra RC, Vriesendorp HM, Andersson BS, Giralt S, Korbling M, Keating MJ, Champlin RE. Allogeneic blood or marrow transplantation for chronic lymphocytic leukaemia: timing of transplantation and potential effect of fludarabine on acute graft-versus-host disease. Br J Haematol. 1997 May;97(2):466-73. doi: 10.1046/j.1365-2141.1997.272673.x. PMID 9163617
- [Background] Rondon G, Giralt S, Huh Y, Khouri I, Andersson B, Andreeff M, Champlin R. Graft-versus-leukemia effect after allogeneic bone marrow transplantation for chronic lymphocytic leukemia. Bone Marrow Transplant. 1996 Sep;18(3):669-72. PMID 8879640
- [Background] van Besien K, Sobocinski KA, Rowlings PA, Murphy SC, Armitage JO, Bishop MR, Chaekal OK, Gale RP, Klein JP, Lazarus HM, McCarthy PL Jr, Raemaekers JM, Reiffers J, Phillips GL, Schattenberg AV, Verdonck LF, Vose JM, Horowitz MM. Allogeneic bone marrow transplantation for low-grade lymphoma. Blood. 1998 Sep 1;92(5):1832-6. PMID 9716615
- [Background] Khouri IF, Keating M, Korbling M, Przepiorka D, Anderlini P, O'Brien S, Giralt S, Ippoliti C, von Wolff B, Gajewski J, Donato M, Claxton D, Ueno N, Andersson B, Gee A, Champlin R. Transplant-lite: induction of graft-versus-malignancy using fludarabine-based nonablative chemotherapy and allogeneic blood progenitor-cell transplantation as treatment for lymphoid malignancies. J Clin Oncol. 1998 Aug;16(8):2817-24. doi: 10.1200/JCO.1998.16.8.2817. PMID 9704734
- [Background] Giralt S, Thall PF, Khouri I, Wang X, Braunschweig I, Ippolitti C, Claxton D, Donato M, Bruton J, Cohen A, Davis M, Andersson BS, Anderlini P, Gajewski J, Kornblau S, Andreeff M, Przepiorka D, Ueno NT, Molldrem J, Champlin R. Melphalan and purine analog-containing preparative regimens: reduced-intensity conditioning for patients with hematologic malignancies undergoing allogeneic progenitor cell transplantation. Blood. 2001 Feb 1;97(3):631-7. doi: 10.1182/blood.v97.3.631. PMID 11157478
- [Background] Slavin S, Nagler A, Naparstek E, Kapelushnik Y, Aker M, Cividalli G, Varadi G, Kirschbaum M, Ackerstein A, Samuel S, Amar A, Brautbar C, Ben-Tal O, Eldor A, Or R. Nonmyeloablative stem cell transplantation and cell therapy as an alternative to conventional bone marrow transplantation with lethal cytoreduction for the treatment of malignant and nonmalignant hematologic diseases. Blood. 1998 Feb 1;91(3):756-63. PMID 9446633